CLINICAL TRIAL: NCT06937216
Title: Evaluation of the Effectiveness of The Volara System Determined by Sputum Movement and Production
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BXU602317; CIV-25-04-052074 (Other: Eudamed)
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Bronchiectasis Adult; COPD
Keywords: Volara; OLE Therapy; mucous clearance
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This study will be a single arm, monocentric, prospective, pilot study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single Group Assignment (Experimental): Each participant will be his/her own control comparing their baseline status to an active treatment period.
  Interventions: Device: Volara therapy

INTERVENTIONS:
Device: Volara therapy — Oscillation and Lung Expansion (OLE) therapy, is a respiratory airway clearance intervention including continuous high-frequency oscillation and continuous positive expiratory pressure

SUMMARY:
The aim of this study is to evaluate the therapeutic effect of therapy with The Volara System on mucus clearance.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the therapeutic effect of therapy with The Volara System on mucus clearance. Mucus volume (mL) measured by Functional Respiratory Imaging (FRI). FRI is a quantitative endpoint that identifies mucus plugs in the segmented airways. Mucus volume will be assessed based on movement of mucus plugs and/or clearance from segmental airways. CT scans are obtained to determine FRI and will be obtained and assessed at baseline and after the 4-week treatment period to assess changes in mucus volume within the airways, associated with the Volara treatment. The study will also provide insight into the mechanism of action of the therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of COPD with or without bronchiectasis.
2. Age ≥ 21 years.
3. Naive to Volara therapy.
4. FEV1 < 80% predicted (based on pulmonary function tests within the past 12 months).
5. Daily sputum production over the prior 2 weeks.
6. Signed informed consent.
7. Stable pulmonary disease defined as no change in disease status.
8. Stable medication regimen for 30 days prior to visit 1, defined as no change in prescribed medications and adherence to their prescribed medications for pulmonary disease

Exclusion Criteria:

1. Anticipated requirement for hospitalisation within the next 35 days (± 1 day).
2. History of pneumothorax within the past 6 months prior to visit 1.
3. History of haemoptysis requiring embolization within the past 12 months prior to visit 1.
4. Inability or unwillingness to perform Volara System therapy as directed, without healthcare provider support.
5. Inability or unwillingness to complete study visits and/or provide follow-up data as required per the study protocol.
6. Inability to complete a 6-minute walk.
7. Actively participating in another clinical trial involving an investigational medication or device.
8. Pregnant females as verified by point of care human chorionic gonadotropin test.
9. Current Intrapulmonary Percussive Ventilation and/or oscillation and lung expansion users.
10. Participant requires a prescribed daily regimen for airway clearance with a device or with manual therapy in addition to Volara.
11. Participant requires mechanical ventilation.
12. Participants with artificial airways

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change in mucus plug volume (mL) | 28 Days
  Assessed based on movement of mucus plugs and/or clearance from segmental airways

CONTACTS AND LOCATIONS:
Locations (1):
- Medimprove, Kontich, Belgium

IPD SHARING:
Plan to Share IPD: No